CLINICAL TRIAL: NCT02252744
Title: Prevalence of Dry Eye Disease in Patients Diagnosed With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Western University of Health Sciences (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Jasmine Yumori, Associate Professor, Western University of Health Sciences
Other Study IDs: WesternU-12irb027
Record Dates: First submitted 2014-09-18; First posted 2014-09-30 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Dry Eye Syndromes; Rheumatoid Arthritis
Keywords: dry eye disease; rheumatoid arthritis
MeSH Terms: conditions — Dry Eye Syndromes; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
This study will evaluate the prevalence of dry eye disease in patients diagnosed with rheumatoid arthritis. No treatment is administered in this study.

DETAILED DESCRIPTION:
We investigated the prevalence of dry eye disease in patients diagnosed with rheumatoid arthritis by information sheets and direct recruitment of patients of potential study participants diagnosed with rheumatoid arthritis. Subjective assessment for dry eye disease was performed using Ocular Surface Disease Index (OSDI) questionnaire. The following objective tests of dry eye disease were employed: tear osmolarity (TO), tear break-up time (TBUT), corneal fluorescein staining score and conjunctival lissamine green staining scores using the National Eye Institute-recommended grading system, and Schirmer without anesthetic. The Dry Eye Severity Grading Scheme highlighted by the Dry Eye WorkShop was adapted to quantify dry eye disease severity level.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis
* 18 years old or older
* Speaks and understands English and/or Spanish

Exclusion Criteria:

* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine W Yumori, OD FAAO, Principal Investigator — Western University of Health Sciences

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- RA Patients: Adult patients diagnosed with rheumatoid arthritis
Period: Overall Study
Arm/Group | RA Patients
Started | 286
Completed | 286
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RA Patients
Number analyzed (Participants) | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.46821 (13.46821)
Gender [Number; unit: participants] — Gender data unavailable for 2 participants
  participants
    Female | 243
    Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 141
  Not Hispanic or Latino | 141
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 22
  White | 216
  More than one race | 0
  Unknown or Not Reported | 22
Region of Enrollment [Number; unit: participants]
  United States | 286

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Diagnosed With Rheumatoid Arthritis Also Found to Have Dry Eye Disease
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | RA Patients
Number analyzed (Participants) | 286
participants | 275

ADVERSE EVENTS:
Arm/Group | RA Patients
Serious Adverse Events (participants affected / at risk) | 0/286
Other Adverse Events (participants affected / at risk) | 0/286

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No